CLINICAL TRIAL: NCT05160480
Title: A Pilot Study of Total-body PET Using FDA-approved Radiotracers Beyond 18F-FDG
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 1837303; EXPLLN21-01 (Other: University of California Davis)
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Breast Cancer; Neuroendocrine Tumors
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total-body PET scan: All participants will receive a dynamic PET scan for up to 90 minutes. This will be followed by two 30 minutes static PET scans at 3 hours +/-20 minutes and 6 hours +/-20 minutes post injection. Subjects injected with 18F-PSMA or 18F-FES will receive a 40 minute scan at 9 hours +/-20 minutes post injection.
  Interventions: Diagnostic Test: Total-body PET imaging

INTERVENTIONS:
Diagnostic Test: Total-body PET imaging — Total-body PET imaging at different timepoints

SUMMARY:
The purpose of this research study is to test new ways to improve the usefulness of the world's first total-body positron emission tomography (PET)/computed tomography (CT) scanner (EXPLORER) by collecting data from PET scans using one of three different imaging agents: 18F-PSMA; 18F-FES; or, 68Ga DOTATATE. These imaging agents are approved by the FDA to be used for patients diagnosed with prostate cancer (18F-PSMA), neuroendocrine tumor (68Ga DOTATATE), or breast cancer (18F-FES).

ELIGIBILITY:
18F-PSMA (n=3) and 68Ga-PSMA (n=3)

Inclusion criteria:

* Persons >18 yo with suspected prostate cancer metastasis
* Prior imaging study (CT, and/or MRI and/or Bone scan and/or Fluciclovine scan) suspicious for metastatic disease, obtained within 4 months from the research scan date.

  68Ga DOTATATE (n=3) or 64Cu-DOTATATE (n=3)

Inclusion Criteria:

* Persons > 18 yo suspicious for or diagnosed with somatostatin receptor positive neuroendocrine tumors (NETs)
* Prior DOTATATE PET/CT scan suspicious for tumor obtained not earlier than 4 months from the research scan date.

Exclusion Criteria:

• Recent administration of long-acting somatostatin analogs

Exclusion Criteria for all participants:

* Adults unable to consent
* Pregnant/lactating persons
* Prisoners
* Unable to lie supine for up to 90 minutes at different timepoints in the PET scanner
* Uncontrolled claustrophobia
* Any significant medical condition that in the opinion of the investigator would prevent the participant from participating and/or adhering to study related procedures or interfere with participant safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by physicians, primary care physicians, radiologists, and research team members who will identify potential participants and notify a research team member to assist with consenting. The research team will also screen potential patients from the oncology clinical schedules. When a potential participant is identified, a member of the research team will contact the referring physician and/or a clinical team member in charge of the patient's care and request permission to contact the patient. If the referring physician/clinical team agrees, a member of the research team will contact the patient.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
measure radiotracer avidity | One study imaging visit lasting up to 10 hours
  measure radiotracer avidity, i.e. standardized uptake value measurements (SUV max and mean) of tumor and normal tissue as a function of time with 18F-PSMA, 18F-FES, 68Ga DOTATATE in a total-body PET scanner among men with suspected prostate cancer metastasis, patients suspicious for or diagnosed with somatostatin receptor positive neuroendocrine tumors, and patients with recurrent or metastatic breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Nardo, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis EXPLORER Molecular Imaging Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No